CLINICAL TRIAL: NCT02625701
Title: Perioperative Fluid Management: Goal-Directed Therapy vs. Restrictive Approach, a Randomized Controlled Trial
Brief Title: Perioperative Fluid Management: Goal-directed Versus Restrictive Strategy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Licker, Professor, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UGeneve - NAC09-022
Record Dates: First submitted 2012-03-22; First posted 2015-12-09 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Complication, Postoperative
Keywords: operative mortality; myocardial infarct, arrhythmia, heart failure, stroke; pneumonia, atelectasis, acute lung injury; surgical site infection; acute kidney injury; body weight
MeSH Terms: conditions — Postoperative Complications; Myocardial Infarction; Arrhythmias, Cardiac; Heart Failure; Stroke; Pneumonia; Pulmonary Atelectasis; Acute Lung Injury; Surgical Wound Infection; Acute Kidney Injury; Body Weight | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients, clinical care givers and assessors are blinded to the the treatment (GDT or restrictive).
  Sealed enveloppes contain the patient' identification number. A person not involved in the study prepare the enveloppes with the identification number.
  Investigators who are assessing the postoperative study outcomes are blinded to the treatment arms
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal-Directed-Therapy (GDT) (Experimental): Besides the basal infusion of crystalloids at 3-6 ml/kg/h, colloids (200 ml) or crystalloids (200 ml) are given over 10 min in the presence of signs of absolute/relative hypovolemia as detected by a fall in cardiac output/stroke volume (CO/SV) or if Pressure Pulse Variation (PVV) or Stroke Volume Variation (SVV) exceeds 10-12%, particularly in the presence. Fluid filling is interrupted when SV fail to increase > 10% (or PVV/SVV =< 10%) Otherwise, vasopressors can be used to achieve appropriate mean arterial pressure (MAP>70 mmHg, within ±20% of baseline).
  Blood losses are replaced with colloids (1:1) or crystalloids (2:1).
  Interventions: Procedure: Goal-directed therapy
- Restrictive strategy (Active Comparator): Crystalloids are given at a fixed rate of 3-6 ml/kg/h. Otherwise, vasopressors can be used to achieve appropriate MAP (>70 mmHg, within ±20% of baseline).
  Blood losses are replaced with colloids (1:1) or crystalloids (2:1). Clinicians in charge of the patients are free to use hemodynamic parameters such as PVV or SVV, always attempting to limit the amount of fluid infusion and to maintain normovolemia
  Interventions: Procedure: Restrictive fluid therapy

INTERVENTIONS:
Procedure: Goal-directed therapy — Optimize CO with additional fluid according to dynamic indices (PPV, SVV, Stroke volume)
  Other Names: GDT
  Arms: Goal-Directed-Therapy (GDT)
Procedure: Restrictive fluid therapy — Keep normovolemia with basal crystalloids infusion (3-6 ml/kg/h) and compensate additional fluid losses with colloids or crystalloids.
  Arms: Restrictive strategy

SUMMARY:
There is no ideal "cookbook recipe" for fluid prescription that would fit every surgical patient.

In this study, the investigators working hypothesis is that the adoption of an integrative algorithm for perioperative fluid and haemodynamic management would improve clinical outcome and reduce hospital resource utilization in noncardiac surgical procedures (major-to-intermediate level of stress.

Two intraoperative fluid strategies will be compared: "Restrictive" vs. "goal-directed therapy (GDT)". In the GDT group, haemodynamic information will be obtained by a flow monitoring device coupled with standard heart rate and blood pressure monitoring.

DETAILED DESCRIPTION:
The rationale of minimizing body weight gain and avoiding unnecessary fluid compensation of the "third compartment" is now well justified and achievement of supra-normal oxygen delivery values is likely not necessary in most surgical patients. Therefore,it would be tempting to adopt fluid restriction protocols given the potentials of better wound healing, faster return of bowel function and shorter hospital stay after major surgical procedures.

Although dynamic flow indices of volume responsiveness have been validated in critically-ill patients, concerns have been raised regarding the risk of overzealous fluid administration in non-critically-ill patients undergoing elective surgery.

To date, RCTs comparing fluid regimen ("liberal" versus "restrictive" or "liberal" versus "GDT") have yielded controversial results with no consensus regarding appropriate fluid administration in the perioperative period. Interestingly, restrictive protocols have been associated with more frequent adverse events (e.g., nausea, vomiting) following minor surgical procedures and concerns have been raised regarding the possibility of tissue hypoperfusion leading to end-organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* elective noncardiac surgery (moderate-high-risk) lasting > 2h hours (, gastrectomy, pancreatectomy, nephrectomy, radical cystectomy, hepatic resection, open colonic or rectal surgery)

Exclusion Criteria:

* end-stage organ failure (hemofiltration/dialysis; Child-Pugh class C or MELD score >22; predicted forced expiratory volume < 30%, severe heart failure)
* life expectancy < 24h
* psychiatric disorders or unability to give independent consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
composite index of serious postoperative adverse events | from date of surgery till hospital discharge or 30-day postoperative
  early postoperative major outcomes: mortality, cardiovascular, respiratory, renal and infectious complications

SECONDARY OUTCOMES:
body weight changes (kg, postoperative value - preoperative value) | from date of surgery till hospital discharge, or 30-day postoperative
  comparison of body weight (preop versus postop value, kg)
fluid balance | intra-operative and first 24hours after surgery
  amount of fluids (ml) infused, amount of fluid losses
  change in body weight
Acute Kidney Injury based on RIFLE | from the day before to 3 days after surgery
  measurements of creatinine (preoperative, postoperative day 1, 2, 3 after surgery) and assessing the changes in glomerular filtration rate (%)
Sequential Organ Failure Assessment (SOFA) | from date of surgery till hospital discharge, up to 15 weeks after date of surgery
  scoring the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems
tissue oximetry (%) | intraoperative period, day of surgery
  Monitoring of oxygen delivery/utilization in the brain area with near-infra-red spectroscopy (NIRS)
survival | survival 1-3 years after surgery
  patients (family, next of kin, doctor) are contacted by phone or mail

CONTACTS AND LOCATIONS:
Overall Officials: Marc Licker, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Department of Anesthesiology, Geneva, Switzerland